CLINICAL TRIAL: NCT05390515
Title: Psoriatic Immune Response to Tildrakizumab
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of California, San Francisco (Other)
Collaborators: Sun Pharmaceutical Industries Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 22-36503
Record Dates: First submitted 2022-05-20; First posted 2022-05-25 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Psoriasis Vulgaris

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Tildrakizumab treatment (Experimental): Biological/vaccine: tildrakizumab
  Interventions: Drug: Tildrakizumab Prefilled Syringe

INTERVENTIONS:
Drug: Tildrakizumab Prefilled Syringe — IL-23 inhibitor

SUMMARY:
This study aims to assess cutaneous and blood immune cell function of patients with psoriasis before and after initiation of treatment with the IL23 blocker, tildrakizumab.

DETAILED DESCRIPTION:
This is a one-arm, open-label study to examine the effect of Tildrakizumab on cutaneous and blood immune cells of psoriatic patients. Ten subjects with moderate to severe psoriasis will be enrolled. Biopsy and blood samples will be collected before and during treatment and undergo molecular profiling to assess for tildrakizumab-corrected signatures.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Patients with moderate-severe psoriasis or > 5% body surface area affected.

Exclusion Criteria:

* taking systemic immunosuppressives in the last 4 weeks
* pregnancy
* severe immunodeficiency (either from genetic or infectious causes).
* tuberculosis or other active serious infection
* active systemic malignancy.
* breast-feeding
* Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in Psoriasis Area and Severity Index (PASI) Score at baseline and 3 months of treatment | Baseline, 3 months
  Change in severity and extent of psoriasis (calculated by Psoriasis Area and Severity Index (PASI) score); scale range of 0 to 72, 72 being maximal disease.

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Cho, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No